CLINICAL TRIAL: NCT04599998
Title: Long-term Follow-up Findings of Inpatients for COVID-19 Pneumonia Related to Lung Functions, Radiology and Exercise Capacity
Brief Title: Long-term Follow-up Findings of Inpatients for COVID-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Koc University Hospital (Other)
Responsible Party: Principal Investigator, Fatma Işıl Uzel, MD, Koc University Hospital
Other Study IDs: 2020.188.IRB1.056
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Covid19
Keywords: Covid19; lung functions; cardiopulmonary exercise testing; thoracic CT; 6 minute walking test; Short form 36 questionnaire
MeSH Terms: conditions — COVID-19 | interventions — Spirometry; Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 inpatients: Patients with laboratory and/or thoracic CT confirmed COVID-19 pneumonia ; older than18 years of age; treated as inpatients; evaluated at 6-12 months after hospital discharge in outpatient clinic
  Interventions: Diagnostic Test: spirometry, thoracic CT, CPET, 6 minute walking test, SF-36 questionnaire

INTERVENTIONS:
Diagnostic Test: spirometry, thoracic CT, CPET, 6 minute walking test, SF-36 questionnaire — Participants will perform spirometry, lung diffusion capacity of carbon monoxide, 6-minute walk test (6MWT), Short form-36 (SF-36) questionnaire and cardiopulmonary exercise testing (CPET) after 6-12 months (Visit 1) of COVID-19. Clinical, laboratory and chest image data during the COVID-19 hospitalization will be obtained from medical records.

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a respiratory tract infection caused by a newly emergent coronavirus (SARS-CoV-2) that can progress to severe multiorgan disease requiring hospitalization. The medium and long-term impact in survivors of COVID-19 on lung function, imaging by thoracic CT, exercise capacity, and health-related quality of life and the relation of these parameters remains to be determined.

DETAILED DESCRIPTION:
Aim: To evaluate medium to late (visit 1: 6-12 months after hospital discharge) effects of COVID-19 on lung function, exercise capacity, thoracic CT findings, symptoms and HRQoL in patients with confirmed diagnosis of SARS-CoV-2 infection and the relation between these parameters.

Material and methods: Prospective cohort of subjects with laboratory and/or thoracic CT confirmed COVID-19 who were treated as inpatients. Participants will perform spirometry, lung diffusion capacity of carbon monoxide, 6-minute walk test (6MWT) and cardiopulmonary exercise testing (CPET) after 6-12 months (Visit 1) of COVID-19. Clinical, laboratory and chest image data during the COVID-19 hospitalization will be obtained from medical records.

The minimum sample size was estimated as 37 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Covid 19 diagnosis
* Ability to read and speak
* Signed informed consent.
* Able to perform exercise testing and walking

Exclusion Criteria:

- Subjects with limited exercise capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Covid-19 diagnosis
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | at 6-12 months after discharge
  in ml
Lung diffusion capacity for carbon monoxide (DLCO) | at 6-12 months after discharge
  DLCO (%predicted); DLCO/alveolar volume- DLCO/VA (%predicted)
6-minute walk test distance | at 6-12 months after discharge
  m
Short-form 36 questionnaire (SF-36) | at 6-12 months after discharge
  scores range between 0 and 100 with higher scores indicating a better HRQoL
Oxygen uptake at peak exercise | at 6-12 months after discharge
  from incremental Cardiopulmonary exercise test (% of predicted)
Minute-ventilation/carbon dioxide output during exercise | at 6-12 months after discharge
  from incremental Cardiopulmonary exercise test (L/L)
Dyspnea during exercise | at 6-12 months after discharge
  from incremental Cardiopulmonary exercise test (measured with 10-point categorical Borg scale
Thoracic CT findings | in the first week of pneumonia and at 6-12 months after discharge
  lung parenchymal abnormalities as percentage of occupied lung
Forced expiratory volume in 1 second | at 6-12 months after discharge
  in ml and %predicted
FEV1/FVC ratio | at 6-12 months after discharge
  in %
Forced vital capacity %predicted (FVC%) | at 6-12 months after discharge
  in %

SECONDARY OUTCOMES:
Signs and symptoms | in the first week of pneumonia and at 6-12 months after discharge
  Recorded separately as present or absent) mortality (recorded as present or absent)
Time to hospital discharge | in hospital
  in days
ICU discharge | in hospital
  in days
Weaning from intubation | in the period of intensive care
  in days
Weaning from supplemental oxygen | in hospital
  in days
Weaning from noninvasive mechanical ventilation | in hospital
  in days
Mortality | in hospital and at 6-12 months after discharge
  recorded as present or absent

CONTACTS AND LOCATIONS:
Overall Officials: Benan Çağlayan, Prof Dr, Study Chair — Koç University Hospital Pulmonology Department
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No